CLINICAL TRIAL: NCT06355648
Title: Advanced Clinical Practitioners in the Emergency Department: a Mixed-method Study of Practice Using Resilient Health Care Principles
Brief Title: Advanced Clinical Practitioners in the ED
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 337181
Record Dates: First submitted 2024-03-18; First posted 2024-04-09 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Healthy Volunteers
Keywords: Advanced Clinical Practitioners; Emergency Department; Resilient Healthcare; Ethnographic; Work-as-done; Work-as-imagined; Resilient Engineering; Socio-technical System; Complex Adaptive Systems
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Emergency Care Advanced Clinical Practitioners: These are nurses, paramedics, or allied health professionals who have undertaken an MSc and work in an Emergency Department.
- Clinical Colleagues of ACPs: These are staff who work directly with ACPs in the ED; they may be doctors, nurses, or allied health professionals.
- Non-Clinical Colleagues: These staff work with Advanced Clinical Practitioners but not in the clinical environment. Examples may be local managers or directors of the organisation.

SUMMARY:
This study is designed to understand better how nurses, paramedics, and other healthcare professionals who have completed extra training to become Emergency Care Advanced Clinical Practitioners (EC-ACPs) work in emergency departments (EDs).

The research questions are:

1) What is the EC-ACP's perception of assimilation into emergency care teams, what tensions are created due to the role, and what system adaptations are required to facilitate integration?

With secondary aims :

1. What are the common organisational factors that affect the implementation of the EC-ACP workforce, and what recommendations can be made to improve Trust-wide implementation?
2. How are EC-ACPs deployed in two contrasting emergency departments, what differences can be identified in their Work-As-Done (WAD), and how does this compare to the Work-As-Imagined (WAI) of the role?

No patient data is being collected; the participants will all be hospital staff:

1. EC-ACP participants will be observed in practice, interviewed, or both.
2. Staff who are not EC-ACPs but work with them will be interviewed for their thoughts on how they work together.

DETAILED DESCRIPTION:
In the UK, a health care role has been developed called Advanced Clinical Practitioners (ACPs). ACPs work in various clinical settings, but this study focuses on those in Emergency Care. While non-medical practitioners have worked in Emergency Departments (EDs) for over 20 years, the ACP role is relatively new. Most ACPs in ED are from a nursing or paramedical background, but they can also be from other allied health professions like physiotherapy. After the base qualification, ACPs undertake a three-year master's degree with clinical portfolios. Once qualified, the goal is to create clinicians who work alongside doctors, seeing, treating, and discharging patients. Unlike previous practitioner roles, EC-ACPs treat the whole spectrum of ED patients, from minor injuries and illnesses to the sickest patients needing the highest level of care.

Observations:

The researcher will aim to shadow x5 EC-ACPs from each site (n=10) for a maximum of five hours each, totalling at least 50 hours of observation in clinical practice. Data collection will aim to capture the variation in how EC-ACPs work by observing EC-ACPs Monday-Sunday between the following hours (08:00-13:00, 13:00-18:00, 18:00-01:00, 01:00-06:00). The researcher will record their observations in the form of field notes, which will be hand-written. Field notes will later be expanded on, typed up, and pseudonymized. During this observation period, researchers may engage in informal discussions with healthcare professionals to clarify what they observe where appropriate, though these will not be audio recorded. Additionally, the researcher will not observe patients while the EC-ACP clinically assesses them. No data will be collected on any patients.

Interviews:

Semi-structured interviews will be undertaken with a range of professional stakeholders (n=20), with ten from each Trust. Interviews will be conducted using an open-ended topic guide, facilitating the exploration of the questions with the participant (Pope & Mays, 2006; Green & Thorogood, 2018). The topic guide will include questions regarding the history of EC-ACP integration into the emergency care team, what specific challenges were encountered, how these were overcome, and what contribution the role has made to the emergency care system from various professional perspectives. If the interview participant was involved in the observation stage of data collection, some questions were asked to clarify observations, deriving more significant insights from the data (Pope & Mays, 2006). Interviews will accommodate the times and dates most suitable for participants. It is envisaged that the 'gatekeepers' at both workplaces will suggest safe and appropriate locations on the two sites for conducting the interviews (Green & Thorogood, 2018). Participants will be informed that interviews will take no more than 45 minutes and will be conducted at an agreeable time. Interview data will be sent to a Kings College London-approved transcription service via secure encrypted email.

Data Analysis:

All formal interview audio recordings will be recorded using a Dictaphone voice recorder with the participant's consent. These recordings will be anonymised and transcribed using a King's College London-approved transcription service. The researcher will personally transcribe 10% of the data interview and observational data to aid familiarisation. Thematic analysis will be conducted to identify recurring themes (Braun and Clarke, 2006). During the coding process, a code book will be created with a list of codes and descriptions to accompany it. The transcripts will be anonymized and uploaded to NVivo to be thematically analysed. The analysis will focus on answering the research questions, using constructs from the conceptual frameworks to sensitize the analysis.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be staff members at the host site.
* ACPs that are observed must work in the Emergency Department.
* All staff must have consented to participate in this research.
* Be over the age of 18.

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will work in an Emergency Department and be selected by identifying their job roles.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-03 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Examine the Work-as-Done of EM-ACPs in Emergency Departments. | 12 months
  Ethnographic data, including observational notes and interview transcripts will be collected and analysed using thematic analysis, underpinned by resilient healthcare theory.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.